CLINICAL TRIAL: NCT05414344
Title: A Randomized Controlled Trial of a Trauma-Informed and Peer-Supported Brief Intervention for Alcohol Users With Interpersonal Trauma
Brief Title: A Brief Intervention for Alcohol Users With Interpersonal Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Principal Investigator, Matthew Woodward, Associate Professor, Western Kentucky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-132
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Heavy Drinking; Alcohol Drinking; Substance Use; Drinking Behavior
Keywords: Brief intervention; Cannabis; Trauma; Alcohol; Drinking; Peer coach
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders; Drinking Behavior; Marijuana Abuse; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either 1) a standard brief intervention 2) a modified brief intervention with peer coaching and trauma-related information or 3) assessment only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Brief Intervention (Experimental): Immediately following completion of the baseline assessment, participants will be texted a link to a secure website which contains the participant's personalized feedback. Personalized feedback is automatically presented via a programming algorithm that is based on the participants baseline survey responses. The personalized feedback component will include a personalized substance use profile, information on peer norms, prior substance-related consequences experienced by the participant, practical costs (e.g., money spent on substances, fees for a DUI), and standard protective behavioral strategies to limit substance-related risk.
  Interventions: Behavioral: Standard Brief Intervention
- Trauma-Informed and Peer-Supported Brief Intervention (TIPS-BI) (Experimental): In addition to the components of the standard brief intervention, the TIPS-BI will include personalized feedback about participants use of substances to cope. Additionally, participants will be provided with psychoeducation about the link between substance use, trauma, and coping motives, and information highlighting the iatrogenic effects that substance use has on negative emotions. Participants will also be given a series of evidence-based alternative coping strategies for managing trauma-related distress such as anxiety, depression, and PTSD. Participants will be asked to set goals related to utilization of these alternative coping strategies. Participants will then be informed that a trained peer who is part of the research team will follow up with them via text message at the monthly time points to review adherence to their goals and offer support.
  Interventions: Behavioral: Trauma-Informed and Peer-Supported Brief Intervention
- Assessment only (Experimental): Following the baseline survey, participants in the assessment only group will be texted again 3 and 6 months later to complete follow up assessments. Following the end of the 6-month follow-up, participants will be offered an opportunity to complete the TIPS-BI without peer coach follow-up.
  Interventions: Behavioral: Assessment only

INTERVENTIONS:
Behavioral: Standard Brief Intervention — Immediately following completion of the baseline assessment, participants will be texted a link to a secure website which contains the participant's personalized feedback. Personalized feedback is automatically presented via a programming algorithm that is based on the participants baseline survey responses. The personalized feedback component will include a personalized substance use profile, information on peer norms, prior substance-related consequences experienced by the participant, practical costs (e.g., money spent on substances, fees for a DUI), and standard protective behavioral strategies to limit substance-related risk.
  Arms: Standard Brief Intervention
Behavioral: Trauma-Informed and Peer-Supported Brief Intervention — In addition to the components of the standard brief intervention, the TIPS-BI will include personalized feedback about participants use of substances to cope. Additionally, participants will be provided with psychoeducation about the link between substance use, trauma, and coping motives, and information highlighting the iatrogenic effects that substance use has on negative emotions. Participants will also be given a series of evidence-based alternative coping strategies for managing trauma-related distress such as anxiety, depression, and PTSD. Participants will be asked to set goals related to utilization of these alternative coping strategies. Participants will then be informed that a trained peer who is part of the research team will follow up with them via text message at the monthly time points to review adherence to their goals and offer support.
  Arms: Trauma-Informed and Peer-Supported Brief Intervention (TIPS-BI)
Behavioral: Assessment only — Following the baseline survey, participants in the assessment only group will be texted again 3 and 6 months later to complete follow up assessments. Following the end of the 6-month follow-up, participants will be offered an opportunity to complete the TIPS-BI without peer coach follow-up.
  Arms: Assessment only

SUMMARY:
The current proposal aims to enhance a mobile-delivered brief intervention for young adults with heavy alcohol use and interpersonal trauma by including adaptive coping strategies for managing trauma-related distress and using peer coaches after delivery of the intervention to maintain treatment gains. Individuals will be randomized to a modified brief intervention incorporating with peer coaches, a standard brief intervention, or assessment only. Participants will be followed up at 3 and 6 months post intervention. The investigators hypothesize that the trauma-informed and peer-supported brief intervention (TIPS-BI) will show low levels of dropout, will be perceived positively by participants, and will result in greater reductions in alcohol use compared to a standard brief intervention and assessment only.

DETAILED DESCRIPTION:
Alcohol is the most frequently used substances in the United States, and emerging adults (EAs) ages 18-25 have the highest rates of heavy substance use of any age group. Heavy and persistent alcohol is linked with a host of negative outcomes in EAs, including poor mental health, lower life satisfaction, cognitive impairments, poor academic performance, increased risk for motor vehicle accidents, and substance use disorders.

Brief interventions (BIs) for substance use typically consist of one to two individual sessions with personalized feedback about substance use. BIs aim to correct inaccurate normative beliefs and highlight personal consequences of substance use. BIs for alcohol use have demonstrated reductions in drinking and alcohol-related problems in numerous clinical trials. However, problems with BIs include 1) effect sizes are typically small and dissipate over time and 2) BIs for substance use demonstrate little to no effectiveness in individuals with interpersonal trauma (i.e., human-perpetrated violence) and interpersonal trauma-related distress. A potential reason for small or null effects of BIs for substance use in EAs are that existing interventions fail to tailor components to specific groups at high risk for substance issues, such as interpersonal trauma survivors. This limited effectiveness may be enhanced by 1) targeting coping motives, a consistent predictor of heavy and persistent alcohol use for interpersonal trauma survivors that is omitted from traditional BIs and 2) use of peer coaches to enhance outcomes following BI delivery.

There are many reasons that greater focus on trauma, coping, and peer influence in BIs could improve outcomes among substance using EAs. Individuals are most likely to experience interpersonal trauma during emerging adulthood, which in turn has been linked to worse mental health, lower social support, and higher rates of alcohol and cannabis use and problems. Studies on alcohol and cannabis use motives suggest that coping with negative emotions are common reasons for substance use among EAs, particularly for EAs with interpersonal trauma, driving heavy use. However, the connections between negative emotions, trauma, substance use, and coping are not addressed in standard BIs. Furthermore, traditional BIs do not provide healthy coping strategies for managing trauma-related negative emotions, despite many empirically supported and adaptive coping strategies that have been identified. Additionally, peer influence has a strong effect on initiation and maintenance of alcohol and cannabis use in EAs, and inclusion of affiliated peers in in-person BIs has been found to enhance treatment efficacy. However, studies have yet to incorporate peers into follow-up of BIs for substance use, despite the demonstrated utility of peer coaches in health interventions for other outcomes (e.g., weight loss).

Importantly, in-person, counselor-delivered BIs have been critiqued as being costly and impractical to implement in real-world settings, inhibiting widespread dissemination. Given that few EAs seek out substance prevention or treatment services, highly accessible, low-cost ways of delivering BIs to this population are needed. Mobile phones are now ubiquitous and represent a particularly advantageous way to provide BIs. Recent research indicates that mobile-delivered substance use interventions show promise in this age group, but given poor treatment engagement often exhibited in many digital health interventions, these approaches may benefit from inclusion of peer coaches following intervention delivery.

The primary goal of the proposed study is to examine the feasibility and efficacy of a mobile-delivered, trauma-informed and peer-supported BI (TIPS-BI) in a sample of EAs with interpersonal trauma histories. The study will enhance and extend research on BIs by: (a) providing intervention content focused on understanding the connection between trauma and substance use and teaching emotion regulation coping skills and (b) incorporating trained peer coaches into text-message-based follow-up. We will conduct a 3-group randomized controlled trial with 165 EAs (ages 18-25; project 60% female) with interpersonal trauma and recent heavy alcohol use. Groups will include Group 1: Mobile-delivered, TIPS-BI with peer coach follow-up (N=55), Group 2: Mobile-delivered standard substance use BI (N=55), and Group 3: Assessment only (N=55)

Aim 1: Examine the feasibility and acceptability of the TIPS-BI. The investigators hypothesize that TIPS-BI will exhibit relatively low levels of dropout (<10%) at follow-up and will be similar to dropout rates shown in the standard BI. The investigators also believe that the TIPS-BI will be perceived by participants as satisfactory, relevant, helpful, and a low burden.

Aims 2 & 3: Evaluate the efficacy of the TIPS-BI in a randomized controlled trial. The investigators hypothesize that the TIPS-BI will be associated with greater reductions in alcohol/cannabis use, alcohol/cannabis problems, and coping motives at 3 and 6-month follow-ups relative to the standard BI and assessment only. The investigators also hypothesize that the TIPS-BI will result in greater increases in coping self-efficacy at 3 and 6-month follow-ups relative to the standard BI and assessment only.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 25
2. Part-time or full-time college student
3. Ability to speak and understand English
4. Access to a cell phone
5. Lifetime history of interpersonal trauma exposure
6. Heavy alcohol use

Exclusion Criteria:

1) Currently receiving psychological therapy or psychotropic medication for substance use.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | Change from Baseline to 3 month follow-up
  The Daily Drinking Questionnaire
Alcohol use | Change from Baseline to 6 month follow-up
  The Daily Drinking Questionnaire
Alcohol use | Change from Baseline to 3 month follow-up
  The Brief Young Adult Alcohol Consequences Questionnaire
Alcohol use | Change from Baseline to 6 month follow-up
  The Brief Young Adult Alcohol Consequences Questionnaire
Cannabis use | Change from baseline to 3-month follow-up
  The Daily Sessions, Frequency, Age of Onset, Quantity of Cannabis Use Inventory (DFAQ-CU)
Cannabis use | Change from baseline to 6-month follow-up
  The Daily Sessions, Frequency, Age of Onset, Quantity of Cannabis Use Inventory (DFAQ-CU)
Cannabis-related problems | Change from baseline to 3-month follow-up
  The Marijuana Problems Scale; scores range from 0-38; higher scores reflect greater problems
Cannabis-related problems | Change from baseline to 6-month follow-up
  The Marijuana Problems Scale; scores range from 0-38; higher scores reflect greater problems
Intervention Feasibility | 6 month follow-up
  Percentage of drop out in the interventions
Intervention Acceptability | 6 month follow-up
  Participants in both the standard and modified brief interventions will be asked to rate on a Likert scale how satisfied they were with the intervention.
Intervention Helpfulness | 6 month follow-up
  Participants in both the standard and modified brief interventions will be asked to rate on a Likert scale how how helpful they found the intervention.

SECONDARY OUTCOMES:
Marijuana use motives | Change from baseline to 3-month follow-up
  The Comprehensive Marijuana Motives Questionnaire; scores range from 3 to 15; higher scores reflect greater endorsement of motives
Marijuana use motives | Change from baseline to 6-month follow-up
  The Comprehensive Marijuana Motives Questionnaire; scores range from 3 to 15; higher scores reflect greater endorsement of motives
Alcohol use motives | Change from baseline to 3-month follow-up
  Modified Drinking Motives Questionnaire - Revised
Alcohol use motives | Change from baseline to 6-month follow-up
  Modified Drinking Motives Questionnaire - Revised
Substance-related coping | Change from baseline to 3-month follow-up
  The Brief Cope Inventory; scores range from 2 to 8; higher scores reflected greater use of the specified coping method
Substance-related coping | Change from baseline to 6-month follow-up
  The Brief Cope Inventory; scores range from 2 to 8; higher scores reflected greater use of the specified coping method
Coping self-efficacy | Change from baseline to 3-month follow-up
  The Coping Self-Efficacy Scale; scores range from 0-260; higher scores reflect greater coping self-efficacy
Coping self-efficacy | Change from baseline to 6-month follow-up
  The Coping Self-Efficacy Scale; scores range from 0-260; higher scores reflect greater coping self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonomo Y, Coffey C, Wolfe R, Lynskey M, Bowes G, Patton G. Adverse outcomes of alcohol use in adolescents. Addiction. 2001 Oct;96(10):1485-96. doi: 10.1046/j.1360-0443.2001.9610148512.x. PMID 11571067
- [Background] Wilk AI, Jensen NM, Havighurst TC. Meta-analysis of randomized control trials addressing brief interventions in heavy alcohol drinkers. J Gen Intern Med. 1997 May;12(5):274-83. doi: 10.1046/j.1525-1497.1997.012005274.x. PMID 9159696
- [Background] Halladay J, Petker T, Fein A, Munn C, MacKillop J. Brief interventions for cannabis use in emerging adults: protocol for a systematic review, meta-analysis, and evidence map. Syst Rev. 2018 Jul 25;7(1):106. doi: 10.1186/s13643-018-0772-z. PMID 30045752
- [Background] Kurtz SP, Pagano ME, Buttram ME, Ungar M. Brief interventions for young adults who use drugs: The moderating effects of resilience and trauma. J Subst Abuse Treat. 2019 Jun;101:18-24. doi: 10.1016/j.jsat.2019.03.009. Epub 2019 Mar 24. PMID 31174710
- [Background] Bountress KE, Cusack SE, Sheerin CM, Hawn S, Dick DM, Kendler KS, Amstadter AB. Alcohol consumption, interpersonal trauma, and drinking to cope with trauma-related distress: An auto-regressive, cross-lagged model. Psychol Addict Behav. 2019 May;33(3):221-231. doi: 10.1037/adb0000457. Epub 2019 Mar 14. PMID 30869917